CLINICAL TRIAL: NCT05668663
Title: Hypovitaminosis C Prevalence and Risk Factors in an Acute Geriatric Unit
Acronym: HYPO-VIT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0883; 2022-A02234-39 (Other: ANSM)
Record Dates: First submitted 2022-12-09; First posted 2022-12-30 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Deficiency, Vitamin C
Keywords: Vitamin C; Hypovitaminosis C; Vitamin C depletion; Vitamin C deficiency; prevalence; risk factors; geriatrics; elderlies; acute care unit
MeSH Terms: conditions — Ascorbic Acid Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elderly patients (Experimental): Only one group of patients will be constituted. It will be composed of 453 patients aged more than 75 years old and hospitalized in a geriatric acute care unit.
  If the patient consent to participate in the study, a 4-mL blood sample will be collected concomitantly with a general laboratory evaluation that will be performed when the patient enters the unit.
  No other sample will be taken., and tThe participation of the patient to the study will end after the result of the test or after the end of the vitamin C supplementation. A telephone call is organized to follow up on any adverse effectswith this blood sample collection.
  No further visit is organised.
  Interventions: Diagnostic Test: Plasmatic Vitamin C concentrations (known as ascorbemia) on a single blood sample

INTERVENTIONS:
Diagnostic Test: Plasmatic Vitamin C concentrations (known as ascorbemia) on a single blood sample — If the patient consents to participate in the study, a 4-mL blood sample will be collected and performed when the patient enters the unit. No other sample will be taken, and the participation of the patient to the study will end after the result of the test or after the end of the vitamin C supplementation. A telephone call is organized to follow up on any adverse effects.
  The blood sample will be collected up to 3 days after admission

SUMMARY:
Vitamin C is essential for numerous biological processes as it acts as a cofactor in various hydroxylation reactions, but also as a powerful antioxidant. As humans have lost the ability to synthetize Vitamin C, this micronutrient is found exclusively in the food, and more particularly in fresh fruits and vegetables.

The term 'hypovitaminosis C' refers to a plasmatic Vitamin C concentration < 28 µmol/L. It encompasses two distinct situations, according to the severity of the deprivation:

* A deeply lowered plasmatic concentration (< 11 µmol/L) is defined as 'Vitamin C deficiency'. The resulting condition is scurvy and its well-known haemorrhagic complications, very likely to be fatal.
* A less low plasmatic concentration (11-27 µmol/L) is defined as 'Vitamin C depletion'. Symptoms are polymorphic and less suggestive, especially for elderly patients. Many studies suggest a chronic Vitamin C depletion may favour the occurrence of various conditions such as cognitive impairment, psychiatric disorders, cardio-vascular diseases, or certain cancers, thereby highlighting the involvement of Vitamin C in many biological processes.

The epidemiology and risk factors of hypovitaminosis C in ageing populations are poorly documented. The few studies dealing with this question are mostly retrospective, including a low number of patients, and relying on an imperfect methodology. Despite these limitations, data suggest hypovitaminosis C could concern up to 50% of the hospitalized geriatric population.

Despite this probably high prevalence, hypovitaminosis C is barely diagnosed and thus rarely supplemented. This is particularly true for the elderlies who are at risk high of being Vitamin C depleted.

Moreover, several risk factors have been described to be associated with Vitamin C depletion or deficiency, sometimes both. But only a few of them have been validated for the geriatric population.

Thus, there is a real need for a better understanding of hypovitaminosis C epidemiology and risk factors in the geriatric population, in order to diagnose earlier, more frequently, and more precisely these cases. It is important to note that an easy and safe supplementation exists (1 g of Vitamin C for 2 weeks).

A better understanding of risk factors is also a key element to apply corrective measures on modifiable risk factors in order to prevent the recurrence of hypovitaminosis C.

In the present research protocol, the investigators hypothesized hypovitaminosis C could concern half of the hospitalized geriatric patients in acute care units.

The primary objective of this study is to evaluate the prevalence of hypovitaminosis C in a geriatric acute care unit, by using a prospective design and including a statistically sufficient number of patients.

The secondary objectives are :

* To determine in this population the prevalence of Vitamin C deficiency,
* To determine in this population the prevalence of Vitamin C depletion,
* To assess the statistical associations between hypovitaminosis C, deficiency, and depletion with already known or pertinent risk factors.
* To follow adverse events with vitamin C supplementation in deficient patients.

ELIGIBILITY:
Inclusion Criteria:

* All patient admitted in the geriatric study acute care unit
* Aged more than 75 years-old.
* Patient able to consent having signed a consent or patient unable to give consent, informed and not opposed to the study to the study and for whom a trustworthy person, or failing that family, or failing that, a close relative, has signed an informed informed consent
* Patient affiliated to a social security system

Exclusion Criteria:

* More than 7 days of hospitalization prior to the admission in the study acute care unit.
* Patients at the end of their life. No biological sample will be collected
* Patients under a "sauvegarde de justice" procedurePatients under legal protection (guardianship, curatorship, "sauvegarde de justice" procedure),
* Patient unable to consent without a trusted person (or family, or close friends) or without a trusted person (or family, or close friend) available within 2 days after the patient's admission.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 434 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Plasmatic Vitamin C concentration (ascorbemia). It is expressed in µmol/L and determined using a laboratory assay. | Day 1 : Ascorbemia will be measured only once for each patient, concomitantly with a general laboratory evaluation that will be performed when the patient enters the unit.
  Ascorbemia will be classified as follows:
  * Normo-ascorbemia for plasmatic concentrations > 28 µmol/L.
  * Hypovitaminosis for plasmatic concentrations < 28 µmol/L

SECONDARY OUTCOMES:
Plasmatic Vitamin C concentration (ascorbemia). It is expressed in µmol/L and determined using a laboratory assay. | Day 1 : Ascorbemia will be measured only once for each patient, concomitantly with a general laboratory evaluation that will be performed when the patient enters the unit.
  For this secondary outcome, hypovitaminosis C will be divided into two sub-groups:
  * Vitamin C deficiency, if the ascorbemia is < 11 µmol/L
  * Vitamin C depletion, if the ascorbemia ranges within 11-27 µmol/L
Risk factors for Hypovitaminosis C | No later than Day 0 : Data are systematically collected during the initial questioning. These data are not specific to the research project.
  Information will be collected about the risk factors of interest for Hypovitaminosis C:
  * Patient identification (age, sex)
  * Medical data (comorbidities, treatments, laboratory data from the general laboratory assessment)
  * Consumption of tobacco or alcohol
  * Life habits and behaviour, autonomy.
Vitamin C depletion | No later than Day 0 : Data are systematically collected during the initial questioning. These data are not specific to the research project.
Vitamin C deficiency | No later than Day 0 : Data are systematically collected during the initial questioning. These data are not specific to the research project.
Follow-up of adverse events in case of vitamin C supplementation. | A call will be made no later than 45 days after the sample is taken for patients supplemented with vitamin C.
  The collection of adverse events from patients supplemented with Vitamin C either by a telephone call from the patient or from the department in which he/she is being treated.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Gériatrique of the Hôpital Edouard Herriot (Pavillon K), Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quillon A, Guittard L, Goldet K, Etienne M, Blond E, Nourredine M, Martin-Gaujard G, Doh S. A cross-sectional study to evaluate hypovitaminosis C prevalence and risk factors in an acute geriatric unit in Lyon, France: the HYPO-VIT-C protocol. BMJ Open. 2023 Aug 23;13(8):e075924. doi: 10.1136/bmjopen-2023-075924. PMID 37612102